CLINICAL TRIAL: NCT03887416
Title: Effect of Dapagliflozin on Nighttime Blood Pressure in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LM Diagnósticos S.L. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAPA-ESR-16-12460; 2017-002125-38 (EudraCT Number)
Record Dates: First submitted 2019-03-08; First posted 2019-03-25 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-03

CONDITIONS: Type2 Diabetes
Keywords: Nighttime blood pressure; Dapagliflozin
MeSH Terms: interventions — dapagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: Type of study: Randomized, multicentric, placebo-controlled, single-blind pilot study.
  Primary Objective: To investigate the effect of the addition of 10 mg daily of dapagliflozin to the treatment of diabetic patients compared to the addition of placebo on the change in nighttime blood pressure (measured by ABPM) over 12 weeks among patients with albuminuria levels ≥ 30 and < 3000 mg/g creatinine and estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): The investigational medicinal product (IMP) is Dapagliflozin 10 MG Oral Tablet [Farxiga] given once daily (film coated tablets, oral use).
  Dapagliflozin 10 MG Oral Tablet [Farxiga] will be administered through out the planned intervention period of the study (12 weeks).
  Dosage form and strength: 10 mg, Green, plain, diamond shaped, film coated tablet (orally)
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet [Farxiga]
- Placebo matching dapagliflozin (Placebo Comparator): The comparator will be placebo oral tablet matching dapagliflozin 10 mg. Placebo will be administered through out the planned intervention period of the study (12 weeks).
  Dosage form and strength: Green, plain, diamond shaped, film coated tablet (orally). Does not contain active ingredient
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10 MG Oral Tablet [Farxiga] — The investigational medicinal product (IMP) is dapagliflozin10 mg given once daily (film coated tablets, oral use).
  Dapagliflozin will be administered through out the planned intervention period of the study (12 weeks).
  Dosage form and strength: 10 mg, Green, plain, diamond shaped, film coated tablet (orally)
  Other Names: Dapagliflozin
  Arms: Dapagliflozin
Drug: Placebo Oral Tablet — The comparator will be placebo oral tablet matching dapagliflozin 10 mg. Placebo will be administered through out the planned intervention period of the study (12 weeks).
  Dosage form and strength: Green, plain, diamond shaped, film coated tablet (orally). Does not contain active ingredient
  Other Names: Placebo
  Arms: Placebo matching dapagliflozin

SUMMARY:
Centres: Three university hospitals and the primary care centres in their area in Madrid (Clínico San Carlos, La Paz, 12 de Octubre) Type of study: Randomized, multicentric, placebo-controlled, single-blind pilot study Main outcome: Nighttime blood pressure in type 2 diabetic patients Objective: To investigate the effect of the addition of 10 mg daily of dapagliflozin to the treatment of diabetic patients compared to the addition of placebo on the change in nighttime blood pressure (measured by ABPM) over 12 weeks among patients withalbuminuria levels ≥ 30 and < 3000 mg/g creatinine and estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2..

Patients: 225 patients with a previous diagnosis of type 2 diabetes and eGFR> 30mL/min x1,73m2, office BP above 140/70 mmHg, HbA1C 7.5-10%, albuminuria levels between 30 mg/g creatinine and 3000 mg/g creatinine and estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2.

Intervention: 10 mg once daily of dapagliflozin or placebo resembling dapagliflozin.

DETAILED DESCRIPTION:
Effect of dapagliflozin on nighttime blood pressure in type 2 diabetes

TYPE OF STUDY: Randomized, multicentric, placebo-controlled, single-blind pilot study.

CENTRES: Three university hospitals and the primary care centres in their area in Madrid (Clínico San Carlos, La Paz, 12 de Octubre)

PRIMARY OBJECTIVE:

To investigate the effect of the addition of 10 mg daily of dapagliflozin to the treatment of diabetic patients compared to the addition of placebo on the change in nighttime blood pressure (measured by ABPM) over 12 weeks among patients with albuminuria levels ≥ 30 and < 3000 mg/g creatinine and estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2.

SECONDARY OBJECTIVES:

* To investigate the effect of the addition of 10 mg daily of dapagliflozin to the treatment of diabetic patients compared to the addition of placebo on the change in nighttime blood pressure (measured by ABPM) over 12 weeks in the subgroup of patients with high (30-300 mg/g creatinine) albuminuria levels.
* To investigate the effect of the addition of 10 mg daily of dapagliflozin to the treatment of diabetic patients compared to the addition of placebo on the change in nighttime blood pressure (measured by ABPM) over 12 weeks in the subgroup of patients with very high (>300 mg/g creatinine) albuminuria levels.
* Changes in albuminuria, office BP and HBA1C in the two subgroups of patients investigated

METHODS:

This clinical trial will be conducted according to this Protocol, under the Regulation (EU) No 536/2014 and all regulatory requirements applicable to clinical trials and following the principles of Good Clinical Practice.

PATIENTS:

Type 2 diabetic patients recruited in the primary care setting in the area of three university hospitals in Madrid, irrespectively of the time since diagnosis and type of treatment received for their diabetes.

DESCRIPTION OF THE INTERVENTION: The drug under evaluation, dapagliflozin, is approved to be used in adults who are 18 or older with type 2 diabetes mellitus for improving glycemic control and can be used in monotherapy when diet and exercise alone do not achieve good glycemic control and metformin use is not indicated due to intolerance, or in combination with other hypoglycemic agents, including insulin, when these, added to diet and exercise do not achieve good glycemic control. In this study it will be used in agreement with the terms in which its use is authorized.

The participants in the study, in addition to the treatment for their diabetes that were receiving from their attending physician, will receive 10 mg once daily of dapagliflozin or placebo resembling dapagliflozinin. The randomization scheme follows below.

RANDOMIZATION:

Two strata will be considered based on albuminuria levels:

* High albuminuria (30-300 mg/g creatinine)
* Very high (>300 mg/g creatinine) Patients will be randomized to either dapagliflozin or placebo in a 2:1 ratio.

Total number of patients: 225; distributed as:

* 150 diabetic patients treated with dapagliflozin (10mg/day in a single dose), half of them with high albuminuria levels (albuminuria 30-300 mg/g of creatinine) and half with very high albuminuria levels (albuminuria > 300 mg/g of creatinine)
* 75 diabetic patients treated with placebo, half of them with high albuminuria levels (albuminuria 30-300 mg/g of creatinine) and half with very high albuminuria levels (albuminuria > 300 mg/g of creatinine) Randomization will be stratified by albuminuria strata and participating hospital (three hospitals); center specific randomization lists (active treatment or placebo) will be prepared centrally at the project office with a treatment code assigned to each patient. Allocation will be concealed by means of sequentially numbered, opaque, sealed envelopes that contain the medication code assigned. The envelopes have to be opened sequentially and only after the participant's name is written on the appropriate envelope.

VISITS, VARIABLES AND MEASUREMENTS:

Four clinical visits are planned in every patient at 0 (recruitment and randomization), 4, 8 and 12 weeks. Information on personal and family history of disease, clinical examination (including office BP determination), ABPM and blood and urine samples will be obtained on visits 0. The variables measured in the blood and urine samples depend on the criterium of the attending physician. For this trial, only HbA1c, serum creatinine, estimated glomerular filtration rate (eGFR) and albuminuria are mandatory. All this information, except personal and family history of disease, will also be collected at week 12. Thirty days after the end of the medication (visit of week 12) all participants will be contacted by telephone to assess safety. For the initial laboratory data required in the CRF, data obtained in primary care in the previous 3 months could be valid. These data will be repeated at the end of the study. Informed consents for the study will be signed by the patients before coming to the hospital. Blood samples extractions included in this protocol will be done, handled and analyzed at each clinical setting according to usual clinical practice. No blood sample storage will be needed in this study.

ABPM will be measured using Mobil-o-Graph that will give us 24 hours brachial and central BP as well as pulse wave velocity and heart rate. As diary of activity of the patient will not be recorded, in this study, nocturnal (or nighttime) blood pressure refers to measurements within the period from 12.00 p.m. to 6.00 a.m.

SAMPLE SIZE CONSIDERATIONS: For the main objective of the study, changes in mean nocturnal systolic blood pressure will be compared between the active treatment and placebo groups.

The use of SGLT2 inhibitors has been reported to be associated with reductions in office blood pressure of 4-8 mmHg, reductions that could be even higher with the use of ambulatory BP monitoring.15 Accepting an alpha error of 0.05 in a two-sided test, 150 patients are needed in the active treatment group and 75 in the placebo group (2:1 randomization) to have an 80% power (beta error=0.2) to detect as statistically significant a difference greater than or equal to 5 mmHg in mean nocturnal BP between placebo and active treatment (conservative estimate of the expected effect). The standard deviation is assumed to be 12 mmHg and it is expected a drop-out rate of 9%.

In the prespecifiedsubgroup analysis by albuminuria levels, this sample size (75 in active treatment and 37 in placebo) allows to detect as statistically significant, within each albuminuria stratum and with the same asumptions and alfa and beta errors, a difference greater than or equal to 7,1 mmHg in the reduction of mean nocturnal BP between both groups (active treatment and placebo), an effect still within what can be expected.

DATA MANAGEMENT: Data will be collected in an electronic CRF by participating doctors and nurses both at the hypertension units and at primary care centers. A range of acceptable values and logical rules among variables will be implemented to improve quality of data and reduce the need of queries.

The processing, communication and transfer of data will be in accordance with the provisions of the Organic Law 15/1999, December 13th, on the protection of personal data.

Trial documentation will be kept and storaged in each site for 25 years after completion of the study.

PLAN OF ANALYSIS: The main analysiswill compare baseline and final visit values of nocturnal blood pressure and all the rest of quantitative variables of interest within each stratum of albuminuria by means of paired t-test. Changes of nighttime blood pressure from baseline to final visit among patients with high and very high albuminuria levels will be compared to placebo with t-test.

Variables will be described by means of mean (and standard deviation) or proportion depending on the type of variable considered. Whenever the test of hypothesis may involve discrete variables, chi-squared testwill be used.

Comparability of treatment and placebo groups will be tested (t-student or chi-squared test, depending on the variable) to assess randomization, and linear regression will be used to adjust for potential confounders, if needed; stratum of albuminuria at randomization will be forced in the model.

To respond to secondary objectives, the same analyses will be done for each stratum of albuminuria at randomization.

Only patients that complete the 3-month follow-up will be analyzed. Patients who do not complete the follow-up will be compared to those who adhere to the protocol.

No interim analysis is planned. A p value<0.05 will be considered as statistically significant.

END OF THE TRIAL:

The trial will end with the last visit of the last patient recruited. The study may be terminated if the study procedures are not being performed according to Good Clinical Practice (GCP). The promotor also may terminate the entire study prematurely if concerns for safety arise within this study or in any other study with dapagliflozin.

ETHICAL ISSUES:

At the recruitment visit, all patients meeting criteria and invited to participate will receive adequate written information on the study and will have the opportunity to ask the investigator any question regarding their participation and will be given enough time to make a decision. Following all this, they will sign and date their acceptance to participate in it prior to randomization. This is a trial proposed as "low level of intervention trial" ["RD 1090/2015 de 4 de diciembre"] and every participant will be covered by an insurance for this instances.

This study will be done conforming to the principles of the Declaration of Helsinki and posterior amendments, Good Clinical Practice and the applicable legislation including the requirements of the Spanish law of data protection ("Reglamento General de Protección de Datos (Reglamento (UE) 2016/679 del Parlamento Europeo y del Consejo, de 27 de abril de 2016", "Ley Orgánica 15/1999 de 13 de diciembre, de protección de datos de carácter personal", and "RD1720/2007"), as described in the "Information for the patient sheet". Data will be entered online and stored securely in a centralized database in a devoted server. To access the eCRF, an user name and password with limited access to allow the development of the study will be assigned to every investigator in the trial (including coordinators and CRO). All personal identification data of the patients will be dissociated from the rest of the data and only the attending physicians will have access to that information to allow the follow-up. All data will be treated anonymously in the analysis and no report from the study will contain any information that allows to identify the patients.

The clinical study will be reviewed by health authorities and an ethic committee and the study will only be started when the approval from the regulatory authorities and the ethic committee is obtained.

At the end of follow-up, every patient will be informed of the treatment group in which he remained during the study and continue the standard care for his/her condition by his/her attending physician.

POTENTIAL RISKS AND BENEFITS OF THE STUDY: The drug under investigation is accepted and of common use in Spain for the treatment of the type of patients that will be included. It will be administered as approved in its specifications. Its use is evidence based and its safety and efficacy are well documented.

All tests and procedures included in the study are normal clinical practice in the diabetic patient with the exception of ABPM that poses no risk for the patient and is basic for the main outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients with a previous diagnosis of type 2 diabetes and

* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min x1.73m2and
* Diagnosis of essential hypertension established at least one year before inclusion visit and suboptimal BP control (office BP above 140/70 mmHg)
* HbA1C 7.5-10%
* Albuminuria levels ≥ 30 mg/g of creatinine

Exclusion Criteria:

* Age < 18 years old or ≥ 75 years old.
* Women of childbearing potential. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Type 1 diabetes
* Albuminuria above 3000 mg/g of creatinine
* Established cardiovascular disease (stable heart failure, peripheral arterial disease or myocardial infarction or stroke within the previous 6 months)
* Intolerance to dapagliflozin
* On treatment with loop diuretic
* On treatment with SGLT2 inhibitors.
* On treatment with pioglitazone.
* Patients diagnosed of hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Patients who routinely work during nightime (period between 11.00 p.m. and 7.00 a.m.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Changes in nighttime blood pressure | 12 weeks
  Changes in mean nighttime blood pressure (systolic and diastolic) between baseline and last visit (units: mmHg)

SECONDARY OUTCOMES:
Changes in office blood pressure. Both systolic and diastolic blood pressure will be assessed | 12 weeks
  Changes in office blood pressure. Both systolic and diastolic blood pressure will be assessed (units: mmHg)
Changes in albuminuria | 12 weeks
  Changes in albuminuria (units:mg/g creatinine)
Changes in HBA1C | 12 weeks
  Changes in HBA1C (units: %)

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Ruilope Urioste, Study Director — Hospital Universitario 12 de Octubre de Madrid
Locations (3):
- Spain (3):
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawes CM, Vander Hoorn S, Rodgers A; International Society of Hypertension. Global burden of blood-pressure-related disease, 2001. Lancet. 2008 May 3;371(9623):1513-8. doi: 10.1016/S0140-6736(08)60655-8. PMID 18456100
- [Background] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Collins R, Peto R, MacMahon S, Hebert P, Fiebach NH, Eberlein KA, Godwin J, Qizilbash N, Taylor JO, Hennekens CH. Blood pressure, stroke, and coronary heart disease. Part 2, Short-term reductions in blood pressure: overview of randomised drug trials in their epidemiological context. Lancet. 1990 Apr 7;335(8693):827-38. doi: 10.1016/0140-6736(90)90944-z. PMID 1969567
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F, Redon J, Dominiczak A, Narkiewicz K, Nilsson PM, Burnier M, Viigimaa M, Ambrosioni E, Caufield M, Coca A, Olsen MH, Schmieder RE, Tsioufis C, van de Borne P, Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S, Clement DL, Coca A, Gillebert TC, Tendera M, Rosei EA, Ambrosioni E, Anker SD, Bauersachs J, Hitij JB, Caulfield M, De Buyzere M, De Geest S, Derumeaux GA, Erdine S, Farsang C, Funck-Brentano C, Gerc V, Germano G, Gielen S, Haller H, Hoes AW, Jordan J, Kahan T, Komajda M, Lovic D, Mahrholdt H, Olsen MH, Ostergren J, Parati G, Perk J, Polonia J, Popescu BA, Reiner Z, Ryden L, Sirenko Y, Stanton A, Struijker-Boudier H, Tsioufis C, van de Borne P, Vlachopoulos C, Volpe M, Wood DA. 2013 ESH/ESC guidelines for the management of arterial hypertension: the Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). Eur Heart J. 2013 Jul;34(28):2159-219. doi: 10.1093/eurheartj/eht151. Epub 2013 Jun 14. No abstract available. PMID 23771844
- [Background] Ruilope LM. Current challenges in the clinical management of hypertension. Nat Rev Cardiol. 2011 Oct 25;9(5):267-75. doi: 10.1038/nrcardio.2011.157. PMID 22027655
- [Background] Ruiz-Hurtado G, Ruilope LM, de la Sierra A, Sarafidis P, de la Cruz JJ, Gorostidi M, Segura J, Vinyoles E, Banegas JR. Association Between High and Very High Albuminuria and Nighttime Blood Pressure: Influence of Diabetes and Chronic Kidney Disease. Diabetes Care. 2016 Oct;39(10):1729-37. doi: 10.2337/dc16-0748. Epub 2016 Aug 11. PMID 27515965
- [Background] Lurbe E, Redon J, Kesani A, Pascual JM, Tacons J, Alvarez V, Batlle D. Increase in nocturnal blood pressure and progression to microalbuminuria in type 1 diabetes. N Engl J Med. 2002 Sep 12;347(11):797-805. doi: 10.1056/NEJMoa013410. PMID 12226150
- [Background] Andrassy KM. Comments on 'KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease'. Kidney Int. 2013 Sep;84(3):622-3. doi: 10.1038/ki.2013.243. No abstract available. PMID 23989362
- [Background] Rajasekeran H, Lytvyn Y, Cherney DZ. Sodium-glucose cotransporter 2 inhibition and cardiovascular risk reduction in patients with type 2 diabetes: the emerging role of natriuresis. Kidney Int. 2016 Mar;89(3):524-6. doi: 10.1016/j.kint.2015.12.038. PMID 26880444
- [Background] Verma S, Garg A, Yan AT, Gupta AK, Al-Omran M, Sabongui A, Teoh H, Mazer CD, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass and Diastolic Function in Individuals With Diabetes: An Important Clue to the EMPA-REG OUTCOME Trial? Diabetes Care. 2016 Dec;39(12):e212-e213. doi: 10.2337/dc16-1312. Epub 2016 Sep 27. No abstract available. PMID 27679584
- [Background] Ferrannini E, Mark M, Mayoux E. CV Protection in the EMPA-REG OUTCOME Trial: A "Thrifty Substrate" Hypothesis. Diabetes Care. 2016 Jul;39(7):1108-14. doi: 10.2337/dc16-0330. PMID 27289126
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Background] Imprialos KP, Sarafidis PA, Karagiannis AI. Sodium-glucose cotransporter-2 inhibitors and blood pressure decrease: a valuable effect of a novel antidiabetic class? J Hypertens. 2015 Nov;33(11):2185-97. doi: 10.1097/HJH.0000000000000719. PMID 26372321
- [Background] Weber MA, Mansfield TA, Cain VA, Iqbal N, Parikh S, Ptaszynska A. Blood pressure and glycaemic effects of dapagliflozin versus placebo in patients with type 2 diabetes on combination antihypertensive therapy: a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Diabetes Endocrinol. 2016 Mar;4(3):211-220. doi: 10.1016/S2213-8587(15)00417-9. Epub 2015 Nov 27. PMID 26620248
- [Background] Parati G, Stergiou G, O'Brien E, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. European Society of Hypertension practice guidelines for ambulatory blood pressure monitoring. J Hypertens. 2014 Jul;32(7):1359-66. doi: 10.1097/HJH.0000000000000221. PMID 24886823
- [Background] Cerezo C, Ruilope LM, Segura J, Garcia-Donaire JA, de la Cruz JJ, Banegas JR, Waeber B, Rabelink TJ, Messerli FH. Microalbuminuria breakthrough under chronic renin-angiotensin-aldosterone system suppression. J Hypertens. 2012 Jan;30(1):204-9. doi: 10.1097/HJH.0b013e32834d9e0f. PMID 22080225
- [Background] Ruiz-Hurtado G, Condezo-Hoyos L, Pulido-Olmo H, Aranguez I, Del Carmen Gonzalez M, Arribas S, Cerezo C, Segura J, Praga M, Fernandez-Alfonso MS, Ruilope LM. Development of albuminuria and enhancement of oxidative stress during chronic renin-angiotensin system suppression. J Hypertens. 2014 Oct;32(10):2082-91; discussion 2091. doi: 10.1097/HJH.0000000000000292. PMID 25033166
- [Background] Pulido-Olmo H, Garcia-Prieto CF, Alvarez-Llamas G, Barderas MG, Vivanco F, Aranguez I, Somoza B, Segura J, Kreutz R, Fernandez-Alfonso MS, Ruilope LM, Ruiz-Hurtado G. Role of matrix metalloproteinase-9 in chronic kidney disease: a new biomarker of resistant albuminuria. Clin Sci (Lond). 2016 Apr 1;130(7):525-38. doi: 10.1042/CS20150517. Epub 2016 Jan 5. PMID 26733721
- [Background] Baldan-Martin M, de la Cuesta F, Alvarez-Llamas G, Gonzalez-Calero L, Ruiz-Hurtado G, Moreno-Luna R, Mourino-Alvarez L, Sastre-Oliva T, Segura J, Padial LR, Vivanco F, Ruilope LM, Barderas MG. Prediction of development and maintenance of high albuminuria during chronic renin-angiotensin suppression by plasma proteomics. Int J Cardiol. 2015 Oct 1;196:170-7. doi: 10.1016/j.ijcard.2015.05.148. Epub 2015 May 29. PMID 26119064
- [Background] Baldan-Martin M, Mourino-Alvarez L, Gonzalez-Calero L, Moreno-Luna R, Sastre-Oliva T, Ruiz-Hurtado G, Segura J, Lopez JA, Vazquez J, Vivanco F, Alvarez-Llamas G, Ruilope LM, de la Cuesta F, Barderas MG. Plasma Molecular Signatures in Hypertensive Patients With Renin-Angiotensin System Suppression: New Predictors of Renal Damage and De Novo Albuminuria Indicators. Hypertension. 2016 Jul;68(1):157-66. doi: 10.1161/HYPERTENSIONAHA.116.07412. Epub 2016 May 23. PMID 27217411
- [Background] de la Cuesta F, Baldan-Martin M, Mourino-Alvarez L, Sastre-Oliva T, Alvarez-Llamas G, Gonzalez-Calero L, Ruiz-Hurtado G, Segura J, Vivanco F, Ruilope LM, Barderas MG. [Cardiovascular risk study in patients with renin-angiotensin system blockade by means of the proteone of circulating extracellular vesicles]. Hipertens Riesgo Vasc. 2016 Jan-Mar;33(1):21-7. doi: 10.1016/j.hipert.2015.07.003. Epub 2015 Sep 19. Spanish. PMID 26826536
- [Background] Wei W, Tolle M, Zidek W, van der Giet M. Validation of the mobil-O-Graph: 24 h-blood pressure measurement device. Blood Press Monit. 2010 Aug;15(4):225-8. doi: 10.1097/MBP.0b013e328338892f. PMID 20216407

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03887416/Prot_SAP_000.pdf